CLINICAL TRIAL: NCT05709782
Title: Phase II Cohort of Spinal Stereotactic Radiotherapy in Patients Using a MR LINAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0589; NCI-2023-00663 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Therapeutic Cohort) (Experimental): Participants in Group 1 will receive spine radiosurgery on the MR LINAC machine, along with imaging scans using the same machine.
  Interventions: Procedure: Spine Radiosurgery; Device: Magnetic Resonance imaging; Radiation: MR-LINAC
- Group 2 (Imaging-only Cohort) (Experimental): Participants in Group 2 will receive spine radiosurgery using a standard radiation therapy machine and have the opportunity to get imaging on the MR LINAC.
  Interventions: Procedure: Spine Radiosurgery; Device: Magnetic Resonance imaging

INTERVENTIONS:
Procedure: Spine Radiosurgery — scan
Device: Magnetic Resonance imaging — scan
Radiation: MR-LINAC — scan
  Arms: Group 1 (Therapeutic Cohort)

SUMMARY:
To learn whether giving spinal stereotactic radiosurgery (SRSS) that uses a more advanced imaging scan method called Magnetic Resonance imaging with a Linear Accelerator (MR-LINAC) during treatment will lead to improved responses to treatment and better quality of life. SRSS is radiation therapy given to the area around your spine.

DETAILED DESCRIPTION:
Primary objective:

• To determine the 6-month local control (LC) of the target site of treatment.

Secondary Objectives:

* To determine the 6-month change in epidural tumor volume (by volumetric measurements where applicable)
* To determine the 1-year local control of the target site

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age ≥ 18 years old
2. Radiographically documented disease of the spine within 4 weeks of registration (candidates with or without epidural disease allowed)
3. Candidate for spine SRS/SBRT as determined by treating Radiation Oncologist or Multidisciplinary Spine Conference review
4. Maximum of 3 contiguous vertebral levels involved with metastasis in the spine to be irradiated allowed
5. Diagnosis of cancer documented
6. Motor strength ≥ 4 out of 5 in the extremity affected by the level of spinal disease planned for radiation
7. Karnofsky Performance score (KPS) ≥ 40 or ECOG score ≤ 3

EXCLUSION CRITERIA:

1. Patients with highly radiosensitive histologies likely to respond to conventional radiation therapy alone (ie lymphoma, multiple myeloma, etc)
2. Patients who are unable to undergo MRI of the spine with contrast
3. Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
M. D. Anderson Symptom Inventory - Spine Tumor (MDASI-SP) questionnaires | through study completion; an average of 1 year
  M. D. Anderson Symptom Inventory - Spine Tumor (MDASI-SP) 0 (symptom has not been present) to 10 (the symptom was as bad as you can imagine it could be) for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Debra N. Yeboa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org